CLINICAL TRIAL: NCT03124862
Title: Accuracy of Acoustic Rainbow Monitoring (ARM) Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TR18351C-TP15637A
Record Dates: First submitted 2017-04-14; First posted 2017-04-24 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Test group (Experimental): The subjects will be enrolled into the test group and will receive ARM sensor.
  Interventions: Device: ARM sensor

INTERVENTIONS:
Device: ARM sensor — Acoustic Monitoring sensor that monitors respiratory rate
  Other Names: RAS-125c

SUMMARY:
The purpose of the study was to conduct a side by side comparison of the accuracy of the respiratory rate (RR) between our Acoustic Rainbow Monitoring (ARM) sensor and the Oridian Microcap Capnograph in healthy adults. Our hypothesis was that the ARM sensor would have comparable or a better performance than the capnograph.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult volunteers

Exclusion Criteria:

* under age of 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-03-17 (Actual); Primary Completion 2012-05-22 (Actual); Study Completion 2012-05-22 (Actual)

PRIMARY OUTCOMES:
Accuracy of Respiratory Rate determination | 40 minutes
  Accuracy is calculated using ARMS analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

IPD SHARING:
Plan to Share IPD: No